CLINICAL TRIAL: NCT01086007
Title: Pain Related Sexual Dysfunction After Laparoscopic Inguinal Hernia Repair
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Innovative Medicines Initiative (Other)
Responsible Party: Principal Investigator, Gitte Linderoth, MD, Rigshospitalet, Denmark
Other Study IDs: H-2-2009-126-B
Record Dates: First submitted 2010-03-11; First posted 2010-03-12 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Sexual Dysfunction; Hernia, Inguinal; Other Chronic Postoperative Pain
Keywords: Groin hernia; chronic pain; Persistent postoperative pain; Laparoscopic inguinal herniotomy; Sexual dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Hernia, Inguinal; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pain patients: Patients with pain related sexual dysfunction after laparoscopic inguinal hernia repair
- Non-pain patients: Patients with no pain related sexual dysfunction after laparoscopic inguinal hernia repair

SUMMARY:
Previous studies have reported that about 3 % of patients who have had open inguinal herniorrhaphy had a visceral, ejaculatory-related pain.

The investigators want to assess this problem among patients after laparoscopic inguinal hernia repair with(self-administered questionnaire study).

ELIGIBILITY:
Inclusion Criteria:

* Male patients
* >18 yrs

Exclusion Criteria:

* Research protection

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who have had a laparoscopic inguinal hernia repair
Sampling Method: Non-Probability Sample
Enrollment: 1172 (Actual)
Dates: Start 2010-02; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gitte Linderoth, MD, Principal Investigator — Section of Surgical Pathophysiology, Rigshospitalet
Locations (1):
- Section of Surgical Pathophysiology, Rigshospitalet, Copenhagen East, Denmark